CLINICAL TRIAL: NCT00201851
Title: Phase III Randomized Study of Immediate Versus Luteal Phase Adjuvant Oophorectomy and Tamoxifen in Premenopausal Women With Hormone Receptor-positive Breast Cancer
Brief Title: Adjuvant Oophorectomy and Tamoxifen in Premenopausal Women With Hormone Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0483
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Asian; Premenopausal; Women; Oophorectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Ovariectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate surgery (Active Comparator): Patient assigned to immediate surgical oophorectomy/mastectomy and Tamoxifen
  Interventions: Drug: Tamoxifen; Procedure: Surgery: Oophorectomy
- Scheduled surgery (Experimental): Patient scheduled for mid-luteal phase surgical oophorectomy/mastectomy plus Tamoxifen
  Interventions: Drug: Tamoxifen; Procedure: Surgery: Oophorectomy
- Immediate Surgery - nonrandomized (Other): Patient in mid-luteal phase at time of enrollment. Assigned to immediate surgical oophorectomy/mastectomy plus Tamoxifen without randomization
  Interventions: Drug: Tamoxifen; Procedure: Surgery: Oophorectomy

INTERVENTIONS:
Drug: Tamoxifen — 20 mg po daily x 5 years
  Other Names: Nolvadex®
Procedure: Surgery: Oophorectomy — Group A-Surgical oophorectomy and mastectomy in estimated 5 days in mid-luteal phase of menstrual cycle (b, c) Group B-Surgical oophorectomy and mastectomy (1-6 days from randomization)(b, c) Group C-Surgical oophorectomy and mastectomy(1-6 days from registration)(c)
  Other Names: ovary removal surgery

SUMMARY:
This trial tests surgical oophorectomy (removal of ovaries) plus Tamoxifen, done at different times in the menstrual cycle, as adjuvant therapy for invasive breast cancer in 510 premenopausal women with Hormone Receptor-positive Breast Cancer. This study is recruiting at hospitals in Philippines, Vietnam, and Morocco.

ELIGIBILITY:
Inclusion Criteria:

* Open for accrual in Asia only
* Female age 18-50,
* premenopausal with regular cycles (>25-35 in length)
* fine-needle aspiration diagnosis
* Stage II-IIIA hormone receptor positive invasive breast cancer
* No prior radiation or chemotherapy
* Must be surgical candidate for bilateral oophorectomy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 740 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Love, M.D., Principal Investigator — International Breast Cancer Research Foundation
Locations (9):
- National Institute of Oncology, Rabat, Morocco
- Philippines (5):
  - Vicente Soto Memorial Medical Center, Cebu
  - East Avenue Medical Center, Manila
  - Philippine General Hospital, Manila
  - Rizal, Manila
  - Santo Toma Hospital, Manila
- Vietnam (3):
  - Danang General, Da Nang
  - Hospital K, National Cancer Institute, Hanoi
  - Hue Central, Huế

REFERENCES:
- [Derived] Hade EM, Young GS, Love RR. Follow up after sample size re-estimation in a breast cancer randomized trial for disease-free survival. Trials. 2019 Aug 23;20(1):527. doi: 10.1186/s13063-019-3632-9. PMID 31443726

RESULTS

PARTICIPANT FLOW:
Groups:
- A - Scheduled Surgery: Patient scheduled for mid-luteal phase surgical oophorectomy/mastectomy plus Tamoxifen
  Tamoxifen: 20 mg po daily x 5 years
  Surgery: Oophorectomy: Group A-Surgical oophorectomy and mastectomy in estimated 5 days in mid-luteal phase of menstrual cycle (b, c) Group B-Surgical oophorectomy and mastectomy (1-6 days from randomization)(b, c) Group C-Surgical oophorectomy and mastectomy(1-6 days from registration)(c)
- B - Immediate Surgery: Patient assigned to immediate surgical oophorectomy/mastectomy and Tamoxifen
  Tamoxifen: 20 mg po daily x 5 years
  Surgery: Oophorectomy: Group A-Surgical oophorectomy and mastectomy in estimated 5 days in mid-luteal phase of menstrual cycle (b, c) Group B-Surgical oophorectomy and mastectomy (1-6 days from randomization)(b, c) Group C-Surgical oophorectomy and mastectomy(1-6 days from registration)(c)
- C- Immediate Surgery - Nonrandomized: Patient in mid-luteal phase at time of enrollment. Assigned to immediate surgical oophorectomy/mastectomy plus Tamoxifen without randomization
  Tamoxifen: 20 mg po daily x 5 years
  Surgery: Oophorectomy: Group A-Surgical oophorectomy and mastectomy in estimated 5 days in mid-luteal phase of menstrual cycle (b, c) Group B-Surgical oophorectomy and mastectomy (1-6 days from randomization)(b, c) Group C-Surgical oophorectomy and mastectomy(1-6 days from registration)(c)
Period: Overall Study
Arm/Group | A - Scheduled Surgery | B - Immediate Surgery | C- Immediate Surgery - Nonrandomized
Started | 252 | 257 | 231
Completed | 244 | 255 | 230
Not Completed | 8 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Ineligible post enrollment | 6 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures were not available on all participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Scheduled Surgery | B - Immediate Surgery | C- Immediate Surgery - Nonrandomized | Total
Number analyzed (Participants) | 244 | 255 | 230 | 729
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (4.5) | 42.3 (4.7) | 42.1 (4.4) | 42.2 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 255 | 230 | 729
  Male | 0 | 0 | 0 | 0
Estrogen receptor status [Number; unit: participants]
  Positive | 226 | 235 | 217 | 678
  Negative | 16 | 19 | 13 | 48
Progesterone receptor status [Number; unit: participants]
  Positive | 218 | 234 | 219 | 671
  Negative | 25 | 20 | 11 | 56
HER2/Neu status [Number; unit: participants]
  Positive | 41 | 45 | 32 | 118
  Negative | 146 | 160 | 153 | 459
Number of positive axillary nodes [Number; unit: participants]
  None | 96 | 111 | 103 | 310
  1-3 | 60 | 73 | 56 | 189
  4+ | 81 | 70 | 68 | 219
Pathologic tumor size [Mean (Standard Deviation); unit: cm] | 4.5 (2.8) | 4.7 (3.2) | 4.1 (2.3) | 4.5 (2.8)
Progesterone level on day of surgery (ng/ml) [Number; unit: participants]
  <2 | 75 | 158 | 74 | 307
  2-4.99 | 27 | 22 | 24 | 73
  5+ | 118 | 57 | 117 | 292

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: 5-year disease-free survival
Time Frame: two- to three-year accrual and initial two or more years of follow-up period
Measure: Number; unit: percentage of participants
Arm/Group | A - Scheduled Surgery | B - Immediate Surgery | C- Immediate Surgery - Nonrandomized
Number analyzed (Participants) | 244 | 255 | 230
percentage of participants | 64 | 71 | 70

ADVERSE EVENTS:
Time Frame: Over entire course of study
Arm/Group | A - Scheduled Surgery | B - Immediate Surgery | C- Immediate Surgery - Nonrandomized
Serious Adverse Events (participants affected / at risk) | 0/244 | 5/255 | 1/230
Other Adverse Events (participants affected / at risk) | 0/244 | 0/255 | 0/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A - Scheduled Surgery (N=244) | B - Immediate Surgery (N=255) | C- Immediate Surgery - Nonrandomized (N=230)
Pregnancy (Reproductive system and breast disorders) | 0 | 1 | 0
Endocervical cancer (Reproductive system and breast disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 1
Nosocomial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No